CLINICAL TRIAL: NCT04160520
Title: Adjuvant Treatment With Pramipexole to Reduce the Dose of Opioids Necessary for Analgesia in Acute Renal Colic
Brief Title: Pramipexole and Morphine for Renal Colic
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECarolinaUniversity
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Renal Colic
Keywords: morphine; Pramipexole; Renal Colic; Kidney Stone; opioids; analgesia; pain relief
MeSH Terms: conditions — Renal Colic; Kidney Calculi; Agnosia | interventions — Pramipexole; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant and study team (i.e. investigators responsible for collecting pain scores) will be blinded as to treatment arm for the duration of the study (2 hours after initiation or until ED discharge/hospital admission). Treatment team (physicians and nurses involved in ED care of the patient) will be unblinded to maintain participant safety and proper medication administration. While the treating physician may be aware of what drugs have been ordered, the need for rescue medications is based on patient pain score at the 30-minute point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pramipexole and half-standard dose of morphine (Experimental): 0.25 mg oral tablet of pramipexole in combination with 0.05mg/kg of IV morphine
  Interventions: Drug: Pramipexole; Drug: Morphine
- Standard dose of morphine and placebo (Active Comparator): 0.1mg/kg of IV morphine in combination with a placebo pill
  Interventions: Drug: Morphine; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Pramipexole — Establish proof of concept that low dose morphine in combination with pramipexole is non-inferior to standard dose morphine with respect to providing analgesia in patients presenting to the ED with pain associated with renal colic.
  Arms: Pramipexole and half-standard dose of morphine
Drug: Morphine — Establish proof of concept that low dose morphine in combination with pramipexole is non-inferior to standard dose morphine with respect to providing analgesia in patients presenting to the ED with pain associated with renal colic.
Drug: Placebo oral tablet — Establish proof of concept that low dose morphine in combination with pramipexole is non-inferior to standard dose morphine with respect to providing analgesia in patients presenting to the ED with pain associated with renal colic.
  Arms: Standard dose of morphine and placebo

SUMMARY:
Opioid analgesics are among the most commonly prescribed class of medications in the US. While opioids may effectively control pain and other sensory disorders under acute conditions, the rates of misuse/abuse and accidental overdose have reached epidemic proportions. Clinicians are being challenged to find alternatives to opioid analgesics, or to reduce their use in treating pain whenever possible. Pre-clinical studies have shown that combining morphine (opioid drug) with pramipexole (dopamine 3 receptor agonist with some D2/D4 action) provides superior analgesia against painful stimuli than morphine alone. This analgesia is maintained even when the dose of morphine is lowered to a dose that is not effective on its own. A recent case report describes the use of this combination to restore pain control in a patient with restless legs syndrome, for which opioids alone have lost their effectiveness (Happe S, Clemens S and Brewer KL, In Review). This application proposes to establish a new therapeutic approach for treatment of a pain associated with renal colic (a common painful condition) using a novel combination of 2 existing, FDA-approved drugs. The immediate goal is to demonstrate that this drug combination can provide similar analgesia to opioid alone, and that analgesia is maintained when the opioid dose is reduced by 50%.

DETAILED DESCRIPTION:
This is a double-blinded randomized controlled trial to take place in the Vidant Medical Center (VMC) Emergency Department (ED). A convenience sample of 96 participants will be drawn from patients presenting to the ED presentation with pain associated with suspected renal colic who do not experience pain relief after initial treatment with nonsteroidal anti-inflammatories.

Written informed consent will be sought by a study team member after screening to ensure all inclusion criteria and no exclusion criteria are met. Once a patient has consented, they will be randomized into 1 of 2 study arms: Arm 1 (Control arm) = 0.1mg/kg of intravenous morphine + placebo pill, single dose Arm 2 (Study arm) = 0.05mg/kg intravenous morphine + 0.25mg pramipexole, single dose. Both arms include a maximum dose of 10mg/kg for the IV morphine. Pain scores will be obtained prior to administration of study drugs, and at 15-minute intervals (+/- 2 mins) after treatment for up to 2 hours, or discharge from the ED. Subjective response to each drug treatment will also be assessed every 15 minutes (+/- 2 mins) after treatment for up to 2 hours, or discharge from ED. Morphine will have a max dose of 10mg IV.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 - 65
* ED presentation with pain associated with suspected renal colic
* Patient reported failure to achieve pain relief with NSAID treatment in ED (additional pain treatment needed per treatment team)

Exclusion Criteria:

* Age < 19 or ≥ 66
* Allergy to any study medication
* Known pregnancy or breastfeeding
* Received opioid prior to enrollment
* Received IV Lidocaine during current ED visit
* Known chronic renal disease
* Currently taking any dopamine receptor agonist or antagonists (Do I need to list?)
* Unable to consent

Ages: 19 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have an effective analgesic response (defined as at least a 50% improvement in pain scores) at 120 minutes post-randomization. | 120 minutes
  Pain scores used are the numerical rating scale (0 low to 10 high) or visual analogue scale (0 low to 100mm high).
Total dose of opioid received at 120 minutes in patients reporting a reduction in pain scores from baseline. | 120 minutes
  Dose of opioid measured in mg/kg
Proportion of patients who require rescue medications at 30 minutes post-randomization. | 30 minutes

SECONDARY OUTCOMES:
Time to reach effective pain reduction (defined as at least a 50% improvement in pain scores) within 120 minutes of treatment. | 120 minutes
  Pain scores used are the numerical rating scale (0 low to 10 high) or visual analogue scale (0 low to 100mm high).
Subjective effects of the drugs measured by scores on the drug effects questionnaire. | 120 minutes
  Drug effects questionnaire rates symptoms from 'not at all' at 0mm to 'extremely' at 100mm.

CONTACTS AND LOCATIONS:
Overall Officials: Kori Brewer, PhD, Principal Investigator — East Carolina University
Locations (1):
- Vidant Medical Center ED, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodgers HM, Yow J, Evans E, Clemens S, Brewer KL. Dopamine D1 and D3 receptor modulators restore morphine analgesia and prevent opioid preference in a model of neuropathic pain. Neuroscience. 2019 May 15;406:376-388. doi: 10.1016/j.neuroscience.2019.03.034. Epub 2019 Mar 23. PMID 30910641
- [Background] Afshar K, Jafari S, Marks AJ, Eftekhari A, MacNeily AE. Nonsteroidal anti-inflammatory drugs (NSAIDs) and non-opioids for acute renal colic. Cochrane Database Syst Rev. 2015 Jun 29;2015(6):CD006027. doi: 10.1002/14651858.CD006027.pub2. PMID 26120804
- [Background] Pathan SA, Mitra B, Bhutta ZA, Qureshi I, Spencer E, Hameed AA, Nadeem S, Tahir R, Anjum S, Cameron PA. A comparative, epidemiological study of acute renal colic presentations to emergency departments in Doha, Qatar, and Melbourne, Australia. Int J Emerg Med. 2018 Jan 3;11(1):1. doi: 10.1186/s12245-017-0160-9. PMID 29299773
- [Background] Patanwala AE, Keim SM, Erstad BL. Intravenous opioids for severe acute pain in the emergency department. Ann Pharmacother. 2010 Nov;44(11):1800-9. doi: 10.1345/aph.1P438. Epub 2010 Oct 26. PMID 20978218
- [Background] Altun A, Yildirim K, Ozdemir E, Bagcivan I, Gursoy S, Durmus N. Attenuation of morphine antinociceptive tolerance by cannabinoid CB1 and CB2 receptor antagonists. J Physiol Sci. 2015 Sep;65(5):407-15. doi: 10.1007/s12576-015-0379-2. Epub 2015 Apr 18. PMID 25894754
- [Background] Altun A, Ozdemir E, Yildirim K, Gursoy S, Durmus N, Bagcivan I. The effects of endocannabinoid receptor agonist anandamide and antagonist rimonabant on opioid analgesia and tolerance in rats. Gen Physiol Biophys. 2015 Oct;34(4):433-40. doi: 10.4149/gpb_2015017. PMID 26374993
- [Background] Terner JM, Barrett AC, Lomas LM, Negus SS, Picker MJ. Influence of low doses of naltrexone on morphine antinociception and morphine tolerance in male and female rats of four strains. Pain. 2006 May;122(1-2):90-101. doi: 10.1016/j.pain.2006.01.019. Epub 2006 Mar 9. PMID 16527399
- [Background] Dourish CT, Hawley D, Iversen SD. Enhancement of morphine analgesia and prevention of morphine tolerance in the rat by the cholecystokinin antagonist L-364,718. Eur J Pharmacol. 1988 Mar 15;147(3):469-72. doi: 10.1016/0014-2999(88)90183-5. PMID 3378566
- [Background] Bijur PE, Schechter C, Esses D, Chang AK, Gallagher EJ. Intravenous bolus of ultra-low-dose naloxone added to morphine does not enhance analgesia in emergency department patients. J Pain. 2006 Feb;7(2):75-81. doi: 10.1016/j.jpain.2005.08.008. PMID 16459272
- [Background] Birnbaum A, Esses D, Bijur PE, Holden L, Gallagher EJ. Randomized double-blind placebo-controlled trial of two intravenous morphine dosages (0.10 mg/kg and 0.15 mg/kg) in emergency department patients with moderate to severe acute pain. Ann Emerg Med. 2007 Apr;49(4):445-53, 453.e1-2. doi: 10.1016/j.annemergmed.2006.06.030. Epub 2006 Sep 15. PMID 16978739
- [Background] Chang AK, Bijur PE, Baccelieri A, Gallagher EJ. Efficacy and safety profile of a single dose of hydromorphone compared with morphine in older adults with acute, severe pain: a prospective, randomized, double-blind clinical trial. Am J Geriatr Pharmacother. 2009 Feb;7(1):1-10. doi: 10.1016/j.amjopharm.2009.02.002. PMID 19281935
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Derived] Girardi C, Duronio J, Patton R, O'Brien K, Clemens S, Brewer KL. A novel opioid/pramipexole combination treatment for the management of acute pain: a pilot study. Front Pain Res (Lausanne). 2024 Sep 24;5:1422298. doi: 10.3389/fpain.2024.1422298. eCollection 2024. PMID 39411383